CLINICAL TRIAL: NCT00084136
Title: Randomized, Open-Label Evaluation of Efficacy of Once-Daily Protease Inhibitor and Once-Daily Non-Nucleoside Reverse Transcriptase Inhibitor-Containing Therapy Combinations for Initial Treatment of HIV-1 Infected Persons From Resource-Limited Settings (PEARLS) Trial
Brief Title: Prospective Evaluation of Anti-retroviral Combinations for Treatment Naive, HIV Infected Persons in Resource-limited Settings
Acronym: PEARLS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5175; 1U01AI068636 (NIH); PEARLS; A5185s; 5K24AI051966-03 (NIH)
Record Dates: First submitted 2004-06-07; First posted 2004-06-08 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Adherence; Drug Resistance; Treatment Failure
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Didanosine; efavirenz; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ZDV/3TC+EFV (Experimental): ZDV/3TC+EFV participants will receive lamivudine/zidovudine and efavirenz
  Interventions: Drug: Efavirenz; Drug: Lamivudine/Zidovudine
- ddI+FTC+ATV (Experimental): ddI+FTC+ATV participants will receive emtricitabine, atazanavir, and enteric-coated didanosine
  Interventions: Drug: Atazanavir; Drug: Didanosine (enteric-coated); Drug: Emtricitabine
- TDF/FTC+EFV (Experimental): TDF/FTC+EFV participants will receive emtricitabine/tenofovir disoproxil fumarate and efavirenz
  Interventions: Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Atazanavir — 400 mg taken orally daily
  Other Names: ATV
  Arms: ddI+FTC+ATV
Drug: Didanosine (enteric-coated) — 400 mg taken orally daily
  Other Names: ddI
  Arms: ddI+FTC+ATV
Drug: Efavirenz — 600 mg taken orally daily
  Other Names: EFV
  Arms: TDF/FTC+EFV; ZDV/3TC+EFV
Drug: Emtricitabine — 200 mg taken orally daily
  Other Names: FTC
  Arms: ddI+FTC+ATV
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200 mg/300 mg taken orally once daily
  Other Names: FTC/TDF
  Arms: TDF/FTC+EFV
Drug: Lamivudine/Zidovudine — 150 mg/300 mg taken orally twice daily
  Other Names: 3TC/ZDV
  Arms: ZDV/3TC+EFV

SUMMARY:
This study compared 3 different three-drug combinations in HIV infected individuals starting their first HIV treatment regimens. Participants were recruited from resource-limited areas in Africa, Asia, South America, Haiti, and also from the United States. The study hypothesis was each of the once daily combinations (PI based, or NNRTI based) would not have inferior efficacy compared to the twice daily NNRTI based combination.

DETAILED DESCRIPTION:
In developed countries, standard effective antiretroviral (ARV) therapy for treatment-naive HIV infected people includes three-drug combinations of two nucleoside reverse transcriptase inhibitors (NRTIs) with either a protease inhibitor (PI) or a non-nucleoside reverse transcriptase inhibitor (NNRTI). However, direct comparisons of ARV efficacy in persons that more closely reflect the worldwide demographics of HIV-1 infection are needed.> > Trial participants were recruited in Africa (Malawi, South Africa, Zimbabwe), Asia (India, Thailand), South America (Brazil, Peru), Haiti, and the United States.>

> All participants were randomly assigned to one of three arms, and random allocation was stratified by 2 factors: country, and screening plasma HIV-1 RNA level (< 100,000 copies/mL versus >= 100,000 copies/mL). Participants assigned to the ZDV/3TC+EFV arm received lamivudine/zidovudine twice daily and efavirenz once daily. Participants assigned to the ddI+FTC+ATV arm received emtricitabine, atazanavir, and enteric-coated didanosine once daily. Participants assigned to the TDF/FTC+EFV arm received emtricitabine, tenofovir disoproxil fumarate, and efavirenz once daily. >

>

> Physical exam and blood collection occurred at entry and at most study visits. Participants experiencing virologic failure were offered a switch to another regimen. >

> On May 23, 2008, the ddI+FTC+ATV was closed following a planned interim review by the study's independent Data and Safety Monitoring Board (DSMB). The DSMB recommendation was based upon compelling evidence that this arm had significantly more virologic failure (and therefore was inferior when) compared to the ZDV/3TC+EFV arm . Participants still receiving ddI+FTC+ATV were offered alternative medications, and all participants continued to be followed. >

> On November 3, 2009, the DSMB recommended that the study close to all follow-up on May 31, 2010, before the designed termination (based on 30% of participants meeting the primary outcome) was met. The board observed that the recent accumulation of primary efficacy events (i.e. regimen failures) was very slow. Therefore, if the study were to continue another 1-2 years, the precision gained for treatment comparisons would likely be small.

ELIGIBILITY:
Inclusion Criteria :>

* HIV-1 infected>
* CD4 count fewer than 300 cells/mm3 >
* Viral load test result>
* Absolute Neutrophil Count at least 750mm3 >
* Hemoglobin at least 7.5 g/dL>
* Platelet count at least 50,000/mm3>
* Calculated creatinine clearance at least 60 mL/min>
* A , A, and alkaline phosphatase <= 5 times upper limit of normal>
* total bilirubin <= 2.5 times upper limit of normal>
* Karnofsky performance score of 70 or higher>
* Plans to stay in the area for the duration of the study>
* Agrees to use acceptable forms of contraception for the duration of the study>

Exclusion Criteria:>

* More than 7 days exposure to ARVs (except for single-dose NVP or ZDV for any period for the purpose of pMTCT)>
* Acute therapy for serious medical illnesses within 14 days prior to study entry>
* Certain abnormal laboratory values>
* Radiation therapy or chemotherapy within 45 days prior to study entry. >
* Any immunomodulator, HIV vaccine, or other investigational therapy within 30 days prior to study entry. >
* Current alcohol or drug abuse that, in the opinion of the site investigator, would interfere with study participation>
* Inflamed pancreas within 3 years prior to study entry>
* Allergy/sensitivity to any of the study drugs or their formulations>
* Heart rate less than 40 beats/min>
* History of untreated, active second- or third-degree heart block>
* Currently detained in jail or for treatment of a psychiatric or physical illness>
* Vomiting or inability to swallow medications>
* Pregnancy>

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1571 (Actual)
Dates: Start 2005-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B. Campbell, MD, Study Chair — University of Colorado, Denver; Timothy Flanigan, MD, Study Chair — The Miriam Hospital; James Hakim, MscClinEpi, FRCP, Study Chair — Department of Medicine, University of Zimbabwe; Nagalingeswaran Kumarasamy, MD, Study Chair — Centre for AIDS Research and Education
Locations (42):
- United States (27):
  - University of Southern California, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Harbor General/UCLA, Torrance, California
  - Univ. of Colorado Health Sciences Center, Denver, Denver, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush-Presbyterian/St. Lukes (Chicago), Chicago, Illinois
  - Cook County Hospital Core Center, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University (St. Louis), St Louis, Missouri
  - HIV Prevention & Treatment CRS, HVTN 722 West 168th Street MSPH Bldg., New York
  - Beth Israel Medical Center, New York, New York
  - Cornell CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Community Health Network, Inc., Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake County Health and Human Services Clinical Research Site, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - University of Texas, Galveston, Galveston, Texas
- Brazil (2):
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Manguinhos, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
- Les Centres GHESKIO CRS, Bicentenaire, Port-au-Prince, Haiti
- India (4):
  - YRG CARE Medical Ctr., VHS Chennai CRS, Rajiv Gandhi Salai Taramani, Chennai
  - NARI Pune CRS, Pune, Maharashtra
  - NARI Clinic at NIV CRS, Maharashtra State, Pune
  - Dr. Kotnis Dispensary, Pune
- Malawi (2):
  - College of Med. JHU CRS, P.O. Box 1131, Blantyre
  - University of North Carolina Lilongwe CRS, Mzimba Road, Lilongwe
- Peru (2):
  - Asociacion Civil Impacta Salud y Educacion - Miraf CRS, Barranco, Lima region
  - San Miguel CRS, San Miguel, Lima region
- South Africa (2):
  - Wits HIV CRS, Johannesburg, Gauteng
  - Durban Adult HIV CRS, Durban, KwaZulu-Natal
- Chiang Mai Univ. ACTG CRS, P.O. Box 80, Chiang Mai, Thailand
- UZ-Parirenyatwa CRS, AIDS Research Unit P.O. Box A178, Harare, Zimbabwe

REFERENCES:
- [Background] Bartlett JA, Johnson J, Herrera G, Sosa N, Rodriguez A, Liao Q, Griffith S, Irlbeck D, Shaefer MS; Clinically Significant Long-Term Antiretroviral Sequential Sequencing Study (CLASS) Team. Long-term results of initial therapy with abacavir and Lamivudine combined with Efavirenz, Amprenavir/Ritonavir, or Stavudine. J Acquir Immune Defic Syndr. 2006 Nov 1;43(3):284-92. doi: 10.1097/01.qai.0000243092.40490.26. PMID 16967040
- [Background] Saag MS. Initiation of antiretroviral therapy: implications of recent findings. Top HIV Med. 2004 Jul-Aug;12(3):83-8. PMID 15310939
- [Background] Tapper ML, Daar ES, Piliero PJ, Smith K, Steinhart C. Strategies for initiating combination antiretroviral therapy. AIDS Patient Care STDS. 2005 Apr;19(4):224-38. doi: 10.1089/apc.2005.19.224. PMID 15857194
- [Derived] Gatechompol S, Zheng L, Bao Y, Avihingsanon A, Kerr SJ, Kumarasamy N, Hakim JG, Maldarelli F, Gorelick RJ, Welker JL, Lifson JD, Hosseinipour MC, Eron JJ, Ruxrungtham K. Prevalence and risk of residual viremia after ART in low- and middle-income countries: A cross-sectional study. Medicine (Baltimore). 2021 Sep 3;100(35):e26817. doi: 10.1097/MD.0000000000026817. PMID 34477118
- [Derived] Firnhaber C, Smeaton LM, Grinsztejn B, Lalloo U, Faesen S, Samaneka W, Infante R, Rana A, Kumarasamy N, Hakim J, Campbell TB. Differences in antiretroviral safety and efficacy by sex in a multinational randomized clinical trial. HIV Clin Trials. 2015 May-Jun;16(3):89-99. doi: 10.1179/1528433614Z.0000000013. Epub 2015 May 15. PMID 25979186
- [Derived] Kantor R, Smeaton L, Vardhanabhuti S, Hudelson SE, Wallis CL, Tripathy S, Morgado MG, Saravanan S, Balakrishnan P, Reitsma M, Hart S, Mellors JW, Halvas E, Grinsztejn B, Hosseinipour MC, Kumwenda J, La Rosa A, Lalloo UG, Lama JR, Rassool M, Santos BR, Supparatpinyo K, Hakim J, Flanigan T, Kumarasamy N, Campbell TB, Eshleman SH; AIDS Clinical Trials Group (ACTG) A5175 Study Team. Pretreatment HIV Drug Resistance and HIV-1 Subtype C Are Independently Associated With Virologic Failure: Results From the Multinational PEARLS (ACTG A5175) Clinical Trial. Clin Infect Dis. 2015 May 15;60(10):1541-9. doi: 10.1093/cid/civ102. Epub 2015 Feb 13. PMID 25681380
- [Derived] Mollan KR, Smurzynski M, Eron JJ, Daar ES, Campbell TB, Sax PE, Gulick RM, Na L, O'Keefe L, Robertson KR, Tierney C. Association between efavirenz as initial therapy for HIV-1 infection and increased risk for suicidal ideation or attempted or completed suicide: an analysis of trial data. Ann Intern Med. 2014 Jul 1;161(1):1-10. doi: 10.7326/M14-0293. PMID 24979445
- [Derived] Campbell TB, Smeaton LM, Kumarasamy N, Flanigan T, Klingman KL, Firnhaber C, Grinsztejn B, Hosseinipour MC, Kumwenda J, Lalloo U, Riviere C, Sanchez J, Melo M, Supparatpinyo K, Tripathy S, Martinez AI, Nair A, Walawander A, Moran L, Chen Y, Snowden W, Rooney JF, Uy J, Schooley RT, De Gruttola V, Hakim JG; PEARLS study team of the ACTG. Efficacy and safety of three antiretroviral regimens for initial treatment of HIV-1: a randomized clinical trial in diverse multinational settings. PLoS Med. 2012;9(8):e1001290. doi: 10.1371/journal.pmed.1001290. Epub 2012 Aug 14. PMID 22936892
- [Derived] Nielsen-Saines K, Komarow L, Cu-Uvin S, Jourdain G, Klingman KL, Shapiro DE, Mofenson L, Moran L, Campbell TB, Hitti J, Fiscus S, Currier J; ACTG 5190/PACTG 1054 Study Team. Infant outcomes after maternal antiretroviral exposure in resource-limited settings. Pediatrics. 2012 Jun;129(6):e1525-32. doi: 10.1542/peds.2011-2340. Epub 2012 May 14. PMID 22585772
- [Derived] Safren SA, Hendriksen ES, Smeaton L, Celentano DD, Hosseinipour MC, Barnett R, Guanira J, Flanigan T, Kumarasamy N, Klingman K, Campbell T. Quality of life among individuals with HIV starting antiretroviral therapy in diverse resource-limited areas of the world. AIDS Behav. 2012 Feb;16(2):266-77. doi: 10.1007/s10461-011-9947-5. PMID 21499794
- [Derived] Firnhaber C, Smeaton L, Saukila N, Flanigan T, Gangakhedkar R, Kumwenda J, La Rosa A, Kumarasamy N, De Gruttola V, Hakim JG, Campbell TB. Comparisons of anemia, thrombocytopenia, and neutropenia at initiation of HIV antiretroviral therapy in Africa, Asia, and the Americas. Int J Infect Dis. 2010 Dec;14(12):e1088-92. doi: 10.1016/j.ijid.2010.08.002. Epub 2010 Oct 18. PMID 20961784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 43 sites from 9 countries: 28 in the US, 4 in India, 2 each in Brazil, Malawi, Peru and South Africa, and 1 each in Haiti, Thailand and Zimbabwe, between May 2005 to August 2007.
Pre-assignment Details: HIV-infected, treatment-naive men and women, at least 18 years of age with CD4+ count <300 cells/mm^3.
Groups:
- ddI+FTC+ATV: ddI+FTC+ATV participants will receive emtricitabine, atazanavir, and enteric-coated didanosine >
  > On May 23, 2008, Arm B was closed following a planned interim review by the study's independent Data and Safety Monitoring Board (DSMB). The DSMB recommendation was based upon compelling evidence that Arm B had significantly more virologic failure (and therefore was inferior when) compared to Arm A. Participants still receiving Arm B medications were offered alternatives, and all participants continued to be followed.
Period: PI Comparison
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Started | 519 | 526 | 0
Completed | 464 (Follow-up was until ddI+FTC+ATV arm was closed per DSMB recommendation on May 23, 2008.) | 479 (Follow-up was until ddI+FTC+ATV arm was closed per DSMB recommendation on May 23, 2008.) | 0
Not Completed | 55 | 47 | 0
Not completed — Death | 10 | 9 | 0
Not completed — Lost to Follow-up | 11 | 8 | 0
Not completed — Withdrawal by Subject | 33 | 30 | 0
Not completed — Clinic site closed | 1 | 0 | 0
Period: NRTI Comparison
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Started | 519 | 0 | 526
Completed | 418 (Follow-up though study closeout period (final visit between April 1 and May 31, 2010).) | 0 | 444 (Follow-up though study closeout period (final visit between April 1 and May 31, 2010).)
Not Completed | 101 | 0 | 82
Not completed — Death | 20 | 0 | 18
Not completed — Lost to Follow-up | 14 | 0 | 12
Not completed — Withdrawal by Subject | 54 | 0 | 38
Not completed — Clinic site closed | 12 | 0 | 14
Not completed — Not reason above | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV | Total
Number analyzed (Participants) | 519 | 526 | 526 | 1571
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9) | 35 (8) | 35 (9) | 35 (9)
Age, Customized [Number; unit: participants]
  Between 18 and 29 years | 141 | 146 | 146 | 433
  Between 30 and 39 years | 244 | 221 | 225 | 690
  Between 40 and 49 years | 100 | 129 | 116 | 345
  At least 50 years | 34 | 30 | 39 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 256 | 242 | 739
  Male | 278 | 270 | 284 | 832
Region of Enrollment [Number; unit: participants]
  Brazil | 79 | 76 | 76 | 231
  Haiti | 35 | 32 | 33 | 100
  India | 81 | 86 | 88 | 255
  Malawi | 74 | 74 | 73 | 221
  Peru | 42 | 48 | 44 | 134
  South Africa | 70 | 70 | 70 | 210
  Thailand | 32 | 33 | 35 | 100
  United States | 70 | 70 | 70 | 210
  Zimbabwe | 36 | 37 | 37 | 110
CD4 count, Continuous [Mean (Standard Deviation); unit: cells/mm^3] — Screening value used for study eligibility as no other pre-randomization CD4 cell counts available
  cells/mm^3 | 163 (85) | 167 (83) | 155 (81) | 162 (83)
CD4 count, Categorical [Number; unit: participants] — Screening CD4 count used for study eligibility as no other pre-randomization counts available.
  participants
    < 50 cells/mm^3 | 68 | 63 | 69 | 200
    Between 50 and 99 cells/mm^3 | 70 | 77 | 82 | 229
    Between 100 and 199 cells/mm^3 | 174 | 161 | 193 | 528
    Between 200 and 249 cells/mm^3 | 104 | 128 | 107 | 339
    Between 250 and 299 cells/mm^3 | 103 | 97 | 75 | 275
Plasma HIV-1 RNA, Continuous [Median (Inter-Quartile Range); unit: log10 copies/mL] | 5.0 [4.6 to 5.4] | 5.1 [4.5 to 5.5] | 5.0 [4.5 to 5.5] | 5.0 [4.6 to 5.5]
Plasma HIV-1 RNA, Categorical [Number; unit: participants]
  <= 400 copies/mL | 3 | 6 | 3 | 12
  Between 400 and 4000 copies/mL | 22 | 19 | 14 | 55
  Between 4001 and 40,000 copies/mL | 103 | 119 | 124 | 346
  Between 40,001 and 400,000 copies/mL | 311 | 283 | 284 | 878
  Between 400,001 and 749,999 copies/mL | 45 | 58 | 55 | 158
  >= 750,000 copies/mL | 35 | 40 | 46 | 121
  Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (PI Comparison)
Description: Time from randomization to the earliest of: scheduled week of first plasma sample meeting virologic failure (two consecutive plasma HIV-1 RNA values 1,000 copies/mL or higher, regardless of whether ARV medications being taken at the time); scheduled week of first AIDS defining diagnosis (WHO Stage 4 (2005), plus microsporidiosis, cyclospora gastroenteritis and Chaga's disease), not attributed to Immune Reconstitution Inflammatory Syndrome (reviewed by chairs); date of death (due to any cause). Plasma drawn every 8 weeks (except confirmation samples could be drawn earlier).
Time Frame: Virologic failure starting 14 weeks following randomization; disease progression starting 12 weeks following randomization; and death occurring at any time following randomization. Follow-up until ddI+FTC+ATV arm closed (May 22, 2008).
Population: ITT (study treatment status and history ignored); censoring time was latest study visit week where plasma HIV-1 RNA was measured.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 526 | 0
weeks
  5th percentile | 16 [16 to 24] | 16 [16 to 16] |
  10th percentile | 40 [24 to 64] | 24 [16 to 32] |
  25th percentile | NA [152 to NA] — Not estimable as the estimate for survival function at all weeks is above 75% | 120 [96 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75% |
Statistical Analysis 1: Comparison: ZDV/3TC+EFV vs ddI+FTC+ATV; Test type: Superiority or Other; p < 0.01, Log Rank — Not adjusted for multiple interim analyses. Peto-Haybittle spending function was used as a basis for calculating the repeated confidence intervals used in interim monitoring; Log-rank test was stratified by country and screening RNA (< 100,000 c/mL vs >= 100,000 copies/mL); Hazard Ratio (HR) = 1.51, 95% CI 2-sided [1.12 to 2.04] — The HR is for ddI+FTC+ATV vs. ZDV/3TC+EFV

2. Primary Outcome: Time to Treatment Failure (NRTI Comparison)
Description: Time from randomization to the earliest of: scheduled week of first plasma sample meeting virologic failure (two consecutive plasma HIV-1 RNA values 1,000 copies/mL or higher, regardless of whether ARV medications being taken at the time); scheduled week of first AIDS defining diagnosis (WHO Stage 4 (2005) plus microsporidiosis, cyclospora gastroenteritis and Chaga's disease), not attributed to Immune Reconstitution Inflammatory Syndrome (reviewed by chairs); date of death (due to any cause). Plasma drawn every 8 weeks (except confirmation samples could be drawn earlier).
Time Frame: Virologic failure starting 14 weeks following randomization; disease progression starting 12 weeks following randomization; and death occurring at any time following randomization. Follow-up through study closure (May 31, 2010).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
weeks
  5th percentile | 16 [16 to 24] |  | 16 [16 to 24]
  10th percentile | 40 [24 to 71] |  | 40 [24 to 64]
  25th percentile | NA [224 to NA] — Not estimable as the estimate for survival function at all weeks is above 75% |  | NA [216 to NA] — Not estimable as the estimate for survival function at all weeks is above 75%
Statistical Analysis 1: Comparison: ZDV/3TC+EFV vs TDF/FTC+EFV; While original study design specified a non-inferiority test, study follow-up stopped early, not due to treatment effect size or futility, but due to slowing accumulation of primary outcome events. Therefore, 2-sided, 95% confidence intervals about the estimated treatment effect (relative effect estimated by a hazard ratio) are provided; Test type: Superiority or Other; Other; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.72 to 1.27] — The HR is for TDF/FTC+EFV vs. ZDV/3TC+EFV

3. Secondary Outcome: Time to Discontinuation of Initial Antiretroviral (ARV) Therapy (PI Comparison)
Description: Time is measured from date of treatment initiation to earliest of the following: date of last participant contact (premature discontinuation of study follow-up); date all ARV medications were held (if all medications held for at least 8 weeks, for any reason); date that any ARV medication was changed (excluding the following single ARV substitutions: stavudine or tenofovir for zidovudine, nevirapine for efavirenz, or didanosine for tenofovir).
Time Frame: Throughout follow-up until ddI+FTC+ATV arm closed (May 22,2008)
Population: Participants not starting study treatment excluded.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 518 | 522 | 0
weeks
  5th percentile | 16 [8 to 22] | 7 [3 to 11] |
  10th percentile | 34 [24 to 46] | 18 [12 to 23] |
  25th percentile | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 75% | 76 [50 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75% |

4. Secondary Outcome: Time to Immunologic Failure (PI Comparison)
Description: Time from randomization to the first scheduled study visit (week 48 or later) with a CD4+ cell count fewer than 100 cells/mm3.
Time Frame: At or after Week 48 (including only follow-up until ddI+FTV+ATV arm closed - May 22,2008)
Population: ITT (ignoring current study treatment status or history)
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 526 | 0
weeks
  1st percentile | 48 [48 to 48] | 48 [48 to 48] |
  5th percentile | 112 [48 to NA] — Not estimable as the upper limit for survival function at all weeks is above 5% | NA [64 to NA] — Not estimable as the estimate for survival function at all weeks is above 5% |

5. Secondary Outcome: Change in CD4 Count From Screening to Weeks 24, 48, 96 (PI Comparison)
Description: Available pre-randomization CD4 cell counts were limited to the single CD4 cell count used for study eligibility (and therefore must have been fewer than 300 cells/mm3).
Time Frame: weeks 24, 48 and 96 (including follow-up until ddI+FTC+ARV arm closed - May 22, 2008)
Population: ITT - ignoring both current treatment status and treatment history.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 526 | 0
cells/mm^3
  Change from screening to week 24 (N=490; N=502) | 112.5 [57.0 to 185.0] | 146.5 [79.0 to 224.0] |
  Change from screening to week 48 (N=474; N=477) | 152.0 [84.0 to 236.0] | 187.0 [111.0 to 272.0] |
  Change from screening to week 96 (N= 188; N=188) | 216.0 [149.0 to 300.5] | 256.0 [142.5 to 371.0] |

6. Secondary Outcome: Time to First Dose Modification or Grade 3 or 4 Adverse Event (PI Comparison)
Description: Time from treatment dispensation to the first occurring of the following: week of first ARV medication change; week of first grade 3 or higher sign/symptom or laboratory abnormality (total bilirubin was excluded) that was at least one grade higher than baseline. Grading used the Division of AIDS (DAIDS) 2004 Severity of Adverse Events Tables.
Time Frame: Throughout study follow-up until ddI+FTC+ATV arm closed (May 22, 2008)
Population: Participants never starting meds excluded. Censoring time is scheduled study week of last clinic visit.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 518 | 522 | 0
weeks
  10th percentile | 4 [4 to 4] | 4 [4 to 8] |
  25th percentile | 12 [12 to 16] | 32 [20 to 40] |
  50th percentile | 96 [72 to 144] | 144 [120 to NA] — Not estimable as the upper limit for survival function at all weeks is above 50% |

7. Secondary Outcome: Plasma HIV-1 Viral Load Fewer Than 400 Copies/ml (PI Comparison)
Description: Number of participants with plasma HIV-1 Viral load fewer than 400 copies/mL at study visit weeks 24 and 48. Closest observed result between 20 and up to 28 weeks (for week 24), and between 44 and up to 52 (for week 48) used if multiple results available. Missing values excluded, and both study treatment status and history ignored.
Time Frame: At Weeks 24 and 48 (including only follow-up until ddI+FTC+ARV arm closed - May 22, 2008)
Population: ITT (ignoring current treatment status or past treatment history); closest value to week 24 (48) used if multiple values available; missing values ignored.
Measure: Number; unit: participants
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 526 | 0
participants
  Week 24: Number with RNA <400 c/mL (N=495; N=506) | 459 | 431 |
  Week 48: Number with RNA <400 c/mL (N=476; N=478) | 437 | 424 |

8. Secondary Outcome: Time to Loss of Virologic Response by Week 48 (Defined by FDA TLOVR Algorithm - Excluding Study Allowed ARV Substitutions)(PI Comparison)
Description: Time from randomization to any of the following events occurring prior to week 48: discontinued ARV regimen (see time to discontinuation of initial ARV therapy above); discontinued study follow-up or died; absence of virologic suppression defined as 2 consecutive plasma HIV-1 RNA values < 400 copies/mL; two consecutive plasma HIV-1 RNA values > 400 copies/mL following virologic suppression.
Time Frame: Week 48 (using follow-up only until closing of ddI+FTV+ATV arm on May 22,2008)
Population: Substitutions not triggering TLOVR event included the following: stavudine or tenofovir-DF for zidovudine; nevirapine for efavirenz; or didanosine for tenofovir-DF.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 526 | 0
weeks
  5th percentile | 0 [0 to 0] | 0 [0 to 0] |
  10th percentile | 16 [8 to 32] | 0 [0 to 0] |
  25th percentile | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 75% | 48 [32 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75% |

9. Secondary Outcome: Time to Loss of Virologic Response at Week 48 (Defined by FDA TLOVR Algorithm - Including All ARV Substitutions)(PI Comparison)
Description: Time from randomization to any of the following events occurring prior to week 48: changed any ARV medication (including permanent discontinuation of all medications); discontinued study follow-up or died; absence of virologic suppression defined as 2 consecutive plasma HIV-1 RNA values < 400 copies/mL; two consecutive plasma HIV-1 RNA values > 400 copies/mL following virologic suppression.
Time Frame: Week 48 (using follow-up only until closing of ddI+FTV+ATV arm on May 22,2008)
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 526 | 0
weeks
  5th percentile | 0 [0 to 0] | 0 [0 to 0] |
  10th percentile | 0 [0 to 0] | 0 [0 to 0] |
  25th percentile | 32 [16 to 48] | 48 [32 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75% |

10. Secondary Outcome: Time to Discontinuation of Initial Antiretroviral (ARV) Therapy (NRTI Comparison)
Description: as for outcome 3
Time Frame: Throughout follow-up until study closed (May 31,2010)
Population: Participants not starting study treatment excluded.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 518 | 0 | 525
weeks
  5th percentile | 16 [8 to 23] |  | 18 [8 to 24]
  10th percentile | 34 [24 to 45] |  | 36 [24 to 48]
  25th percentile | 163 [120 to 200] |  | 201 [160 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75%

11. Secondary Outcome: Time to Immunologic Failure (NRTI Comparison)
Description: as for outcome 4
Time Frame: At or after Week 48 (including all follow-up through study closure - May 31,2010)
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
weeks
  1st percentile | 48 [48 to 48] |  | 48 [48 to 48]
  5th percentile | 128 [48 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95% |  | 104 [48 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95%
  10th percentile | NA [248 to NA] — Not estimable as the estimates for survival function at all weeks is above 90% |  | NA [NA to NA] — Not estimable as all estimates for survival function at all weeks is above 90%

12. Secondary Outcome: Change in CD4 Count From Screening to Weeks 24, 48, 96 (NRTI Comparison)
Description: as for outcome 5
Time Frame: weeks 24, 48 and 96 (including all follow-up through to study closure on May 31, 2010)
Population: ITT - ignoring both current treatment status and treatment history.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
cells/mm^3
  Change from screening to week 24 (N=490; N=498) | 112.5 [57 to 185] |  | 120.5 [67 to 181]
  Change from screening to week 48 (N=480; N=485) | 151.5 [84 to 233.5] |  | 159 [97 to 237]
  Change from screening to week 96 (N=458; N=471) | 220.5 [143 to 313] |  | 226 [142 to 321]

13. Secondary Outcome: Plasma HIV-1 Viral Load Fewer Than 400 Copies/ml (NRTI Comparison)
Description: as for outcome 7
Time Frame: At Weeks 24 and 48 (including follow-up through to study closure on May 31, 2010)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
participants
  Week 24: Number with RNA <400 c/mL (N=495; N=500) | 459 |  | 448
  Week 48: Number with RNA <400 c/mL (N=482; N=487) | 442 |  | 455

14. Secondary Outcome: Time to Loss of Virologic Response at Week 48 (Defined by FDA TLOVR Algorithm - Excluding Study Allowed ARV Substitutions)(NRTI Comparison)
Description: as for outcome 8
Time Frame: Week 48 (using follow-up through study closure on May 31,2010)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
weeks
  5th percentile | 0 [0 to 0] |  | 0 [0 to 0]
  10th percentile | 16 [0 to 32] |  | 24 [0 to 32]

15. Secondary Outcome: Time to Loss of Virologic Response at Week 96 (Defined by FDA TLOVR Algorithm - Excluding Study Allowed ARV Substitutions)(NRTI Comparison)
Description: Time from randomization to any of the following events occurring prior to week 96: discontinued ARV regimen (see time to discontinuation of initial ARV therapy above); discontinued study follow-up or died; absence of virologic suppression defined as 2 consecutive plasma HIV-1 RNA values < 400 copies/mL; two consecutive plasma HIV-1 RNA values > 400 copies/mL following virologic suppression.
Time Frame: Week 96 (using follow-up through to study closure on May 31,2010)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
weeks
  5th percentile | 0 [0 to 0] |  | 0 [0 to 0]
  10th percentile | 16 [0 to 32] |  | 24 [0 to 32]
  25th percentile | NA [88 to NA] — Not estimable as the estimates for survival function at all weeks is above 75% |  | NA [NA to NA] — Not estimable as all estimates for survival function at all weeks is above 75%

16. Secondary Outcome: Time to Loss of Virologic Response at Week 48 (Defined by FDA TLOVR Algorithm - Including All ARV Substitutions)(NRTI Comparison)
Description: as for outcome 9
Time Frame: Week 48 using follow-up through study closure on May 31,2010
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
weeks
  5th percentile | 0 [0 to 0] |  | 0 [0 to 0]
  10th percentile | 0 [0 to 0] |  | 0 [0 to 24]
  25th percentile | 32 [16 to 48] |  | NA [NA to NA] — Not estimable as all estimates for survival function at all weeks is above 75%

17. Secondary Outcome: Time to Loss of Virologic Response at Week 96 (Defined by FDA TLOVR Algorithm - Including All ARV Substitutions)(NRTI Comparison)
Description: Time to any of the following events occurring prior to week 96: changed any ARV medication (including permanent discontinuation of all medications); discontinued study follow-up or died; absence of virologic suppression defined as 2 consecutive plasma HIV-1 RNA values < 400 copies/mL; two consecutive plasma HIV-1 RNA values > 400 copies/mL following virologic suppression.
Time Frame: Week 96 using follow-up through study closure on May 31,2010
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 519 | 0 | 526
weeks
  5th percentile | 0 [0 to 0] |  | 0 [0 to 0]
  10th percentile | 0 [0 to 0] |  | 0 [0 to 24]
  25th percentile | 32 [16 to 56] |  | NA [80 to NA] — Not estimable as the estimates for survival function at all weeks is above 75%

18. Secondary Outcome: Time to First Dose Modification or Grade 3 or 4 Adverse Event (NRTI Comparison)
Description: as for outcome 6
Time Frame: Throughout study follow-up until study closure (May 31, 2010)
Population: Participants never starting meds excluded. Censoring time is scheduled study week of last clinic visit.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Number analyzed (Participants) | 518 | 0 | 525
weeks
  10th percentile | 4 [4 to 4] |  | 4 [4 to 8]
  25th percentile | 12 [12 to 16] |  | 32 [24 to 48]
  50th percentile | 112 [72 to 136] |  | 224 [192 to NA] — Not estimable as the upper limit for survival function at all weeks is above 50%

ADVERSE EVENTS:
Time Frame: Throughout study follow-up (until May 31, 2010 or earlier only if participant prematurely left the study).
Description: Standard Level reporting by DAIDS EAE Manual,May 6, 2004(http://rcc.tech-res.com/safetyandpharmacovigilance/). ATV-related, asymptomatic hyperbilirubinemia or jaundice without LFT elevation does not require (EAE) reporting. IRIS events do not fulfill the DAIDS EAE reporting criteria, even if the event is severe in intensity.
Arm/Group | ZDV/3TC+EFV | ddI+FTC+ATV | TDF/FTC+EFV
Serious Adverse Events (participants affected / at risk) | 86/519 | 84/526 | 55/526
Other Adverse Events (participants affected / at risk) | 481/519 | 521/526 | 489/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZDV/3TC+EFV (N=519) | ddI+FTC+ATV (N=526) | TDF/FTC+EFV (N=526)
Anaemia (Blood and lymphatic system disorders) | 12 | 2 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 17 | 8 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 5 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 4 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 4 | 5 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 8 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
AIDS related complex (Infections and infestations) | 1 | 0 | 0
Abortion infected (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Chikungunya virus infection (Infections and infestations) | 1 | 0 | 0
Corynebacterium sepsis (Infections and infestations) | 0 | 1 | 0
Cryptococcosis (Infections and infestations) | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 2
Encephalitis viral (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 4 | 1
HIV infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Malaria (Infections and infestations) | 0 | 1 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 8 | 2
Blood creatine increased (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 2 | 3 | 2
Neutrophil count decreased (Investigations) | 5 | 4 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 2 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 | 5 | 2
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 3
Suicide attempt (Psychiatric disorders) | 1 | 2 | 5
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Dapsone syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZDV/3TC+EFV (N=519) | ddI+FTC+ATV (N=526) | TDF/FTC+EFV (N=526)
Lymphadenopathy (Blood and lymphatic system disorders) | 27 | 24 | 30
Ocular icterus (Eye disorders) | 7 | 49 | 12
Abdominal pain (Gastrointestinal disorders) | 39 | 57 | 52
Diarrhoea (Gastrointestinal disorders) | 43 | 46 | 63
Nausea (Gastrointestinal disorders) | 48 | 44 | 36
Vomiting (Gastrointestinal disorders) | 60 | 47 | 50
Chest pain (General disorders) | 34 | 37 | 28
Pain (General disorders) | 36 | 43 | 42
Pyrexia (General disorders) | 96 | 120 | 112
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 34 | 6
Herpes zoster (Infections and infestations) | 38 | 41 | 33
Malaria (Infections and infestations) | 43 | 44 | 40
Oral candidiasis (Infections and infestations) | 24 | 23 | 27
Pharyngitis (Infections and infestations) | 19 | 20 | 28
Pneumonia bacterial (Infections and infestations) | 28 | 30 | 28
Upper respiratory tract infection (Infections and infestations) | 37 | 37 | 45
Alanine aminotransferase increased (Investigations) | 220 | 261 | 265
Aspartate aminotransferase increased (Investigations) | 269 | 304 | 289
Blood albumin abnormal (Investigations) | 174 | 188 | 188
Blood alkaline phosphatase increased (Investigations) | 18 | 37 | 24
Blood bicarbonate abnormal (Investigations) | 35 | 60 | 48
Blood bilirubin increased (Investigations) | 44 | 397 | 39
Blood phosphorus decreased (Investigations) | 75 | 87 | 80
Blood potassium decreased (Investigations) | 30 | 29 | 39
Blood sodium decreased (Investigations) | 72 | 94 | 69
Haemoglobin decreased (Investigations) | 88 | 90 | 79
Lipase increased (Investigations) | 16 | 56 | 11
Neutrophil count decreased (Investigations) | 114 | 93 | 103
Platelet count decreased (Investigations) | 45 | 36 | 52
Weight decreased (Investigations) | 33 | 20 | 28
White blood cell count decreased (Investigations) | 35 | 41 | 52
Decreased appetite (Metabolism and nutrition disorders) | 26 | 22 | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 36 | 25
Decreased vibratory sense (Nervous system disorders) | 12 | 30 | 23
Dizziness (Nervous system disorders) | 49 | 29 | 29
Headache (Nervous system disorders) | 78 | 90 | 91
Hypoaesthesia (Nervous system disorders) | 24 | 21 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 27 | 24
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 20 | 30 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 81 | 97 | 106
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 28 | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 | 27 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 39 | 31
Productive cough (Respiratory, thoracic and mediastinal disorders) | 26 | 26 | 22
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 38 | 44 | 57
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 38 | 25
Rash (Skin and subcutaneous tissue disorders) | 33 | 38 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights